CLINICAL TRIAL: NCT02991989
Title: Does Exercise Snacking Improve Muscle Function in Older Adults?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Mr Oliver Perkin, Principle Investigator, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UoB-ESS-01
Record Dates: First submitted 2016-12-06; First posted 2016-12-14 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Muscle Function
Keywords: Home-based exercise; Exercise snacking; Protein; Yogurt
MeSH Terms: interventions — Yogurt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Snacking Group (Experimental): For 28 days, this group will be asked to perform two 'exercise snacks' a day; once in the morning and once in the evening. They will also be asked to consume 150 g of yogurt with the breakfast meal. The yogurt will be provided by the researchers.
  Interventions: Behavioral: Exercise Snacking; Dietary Supplement: Yogurt
- Yogurt Only Group (Other): For 28 days, this group will be asked to consume 150 g of yogurt with the breakfast meal. The yogurt will be provided by the researchers. Apart from consuming the yogurt, this group will be asked to continue their normal lifestyle.
  Interventions: Dietary Supplement: Yogurt

INTERVENTIONS:
Behavioral: Exercise Snacking — Each bout of exercise snacking consists of 5 exercise. Each exercise is performed for one minute, with aim of completing as many repetitions as possible of that exercise in that minute. One minute of rest is observed between each exercise of the exercise snack. The five exercises are; sit-to-stand from a chair, marching on the spot, seated knee extensions alternating legs, standing knee bends alternating legs, and standing calf raises. The sit-to-stand exercise is always performed first, with the number of repetitions achieved recorded, and subsequent exercises performed in any order without recording of repetitions.
  Two exercise snacks are completed each day for 28 days; once in the morning and once in the evening, or at least separated by 2 hours.
  Arms: Exercise Snacking Group
Dietary Supplement: Yogurt — Participants are asked to consume 150 g of yogurt (Arla, Skyr- natural flavour) with their breakfast meal. Participants may substitute the yogurt for another part of their regular breakfast, or add the yogurt to their regular breakfast, with participants asked to record a log book of daily yogurt consumption and to complete a three day food diary during the last week of the 28 day intervention period.

SUMMARY:
Muscle size declines at around 0.5-1% per year after 50 years of age, with muscle strength declining up to twice as fast as muscle size. This may eventually lead to loss of independence if tasks of daily living become too strenuous to be performed safely. Exercise is recognized as a safe and effective means to counteract muscle loss during aging, however access to gym equipment may be logistically challenging or unpalatable to older adults. This research is designed to investigate the effect of 28 days of home-based leg exercise that doesn't require exercise equipment or supervision (exercise snacking), accompanied with a daily protein supplement in the form of commercially available yogurt, on the skeletal muscle health (i.e. function and size) of independent, community-dwelling older adults. To achieve this, two groups will be compared; one group will undertake exercise snacking and consume a 150 g yogurt with the breakfast meal for four weeks, with the second group only receiving the daily yogurt with no exercise snacking.

DETAILED DESCRIPTION:
The study will require potential participants to undergo an eligibility screening with a member of the research team, followed by a period of seven days of habitual activity monitoring and 3 days of diet recording. Eligible participants will be allocated into study groups by way of minimization based on sex, age, BMI, and number of sit-to-stands performed in a minute. Participants will undertake two familiarisation sessions with strength, power, neural drive, and balance tests at least seven days apart, the first following eligibility screening and the second familiarisation session at least five days before the first main trial.

Thereafter, both groups will undertake a main trial the day before commencing 28 days of daily 150 g yoghurt supplement with the breakfast meal, with the exercise snacking group (ES) also undertaking two bouts of exercise snacking a day. The main trial will include measures of leg muscle function and neural drive, standing and single leg balance, and movement co-ordination during tasks of everyday ambulation. Participants will wear a physical activity monitor and pedometer for the seven days and record diet for three days during the last week of the intervention. The day after the intervention period, a follow-up main trial will be conducted as per the first main trial, followed by an optional qualitative interview regarding participant's experience of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Not underweight or obese (body mass index ≥20 and ≤ 30 kg/m2)
* Not regularly engaging in recreational sports or structured exercise (once a week or more).
* Non-smoker (for >5 years)
* Healthy (see exclusion criteria)

Exclusion Criteria:

* Any chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, peripheral arterial disease, insulin- or non-insulin dependent diabetes or other metabolic disorders - all ascertained through preliminary screening.
* Individuals with a history of bone, joint or neuromuscular problems or a current musculoskeletal injury ascertained through preliminary screening.
* Individuals with any joint replacement surgical implants or other artifacts containing metal.
* Individuals with a clinically diagnosed allergy or intolerance of dairy products.
* Individuals with contraindications to exercise including chest pain, dizziness, or loss of consciousness, or who have been instructed by their doctor to only do physical activity recommended by them.
* Individuals who score less than 8 on the Short Physical Performance Battery or score zero on any component of the test.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-20 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
60 second sit to stand test | 28 days- change from pre- to post- intervention period
  The participant is asked to stand up from sitting in a chair whilst keeping their arms folded across their chest, then return to the seated position as many times as possible in a minute.

SECONDARY OUTCOMES:
Lower limb muscle power | 28 days- change from pre- to post- intervention period
  Measured during leg pressing
Lower limb movement outcome variability | 28 days- change from pre- to post- intervention period
  Measured during leg pressing
Lower limb muscle cross-sectional area | 28 days- change from pre- to post- intervention period
  Measured using peripheral quantitative computed tomography at 66% distal calf length and 25% and 50% distal thigh length
Lower limb muscle cross-sectional tissue density | 28 days- change from pre- to post- intervention period
  Measured using peripheral quantitative computed tomography at 66% distal calf length and 25% and 50% distal thigh length
Body composition | 28 days- change from pre- to post- intervention period
  Measured using Dual Energy X-ray Absorptiometry
Gastrocnemius and quadriceps muscle fibre pennation angle | 28 days- change from pre- to post- intervention period
  Measured using ultrasonography at 66% distal length of calf length and 50% distal thigh length
Gastrocnemius and quadriceps muscle fibre length | 28 days- change from pre- to post- intervention period
  Measured using ultrasonography at 66% distal length of calf length and 50% distal thigh length
Postural sway during standing balance with eyes open and closed | 28 days- change from pre- to post- intervention period
  Measured using a force plate
Single leg balance | 28 days- change from pre- to post- intervention period
  Measured using the Y-balance test
Six minute walk test | 28 days- change from pre- to post- intervention period
  The participant will be asked to walk as many times between two cones places 15 meters apart as possible in six minutes.
Movement co-ordination during walking and sit to stands | 28 days- change from pre- to post- intervention period
  Measured by Qualisys motion capture and force plates
Central drive of the plantar flexors | 28 days- change from pre- to post- intervention period
  Measured through the interpolated twitch technique

CONTACTS AND LOCATIONS:
Overall Officials: Keith Stokes, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers